CLINICAL TRIAL: NCT02525042
Title: Study of the Genetic Susceptibility to Ankylosing Spondylitis by Functional Genomics Approach
Brief Title: Genetic Susceptibility to Ankylosing Spondylitis (AS) by Functional Genomics Approach
Acronym: GENOSPA
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI09031
Record Dates: First submitted 2015-08-03; First posted 2015-08-17 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-06

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing Spondylitis; Dendritic cells (DC); RNA; Axial spondyloarthritis; Lod score; Human leucocyte antigen (HLA-B27)
MeSH Terms: conditions — Spondylitis, Ankylosing; Axial Spondyloarthritis

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — RNA is extracted from cells obtained from blood samples (leukocytes).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients with ankylosing spondylitis: Patients with ankylosing spondylitis
- Comparator 1: family controls
- Comparator 2: population controls

SUMMARY:
The main objective is to identify in the candidate regions of differentially expressed genes by comparing the transcriptome of dendritic cells derived from circulating monocytes between cases and controls. Cases and family controls will be matched on the presence of HLA-B27 and depending on haplotype association studies to correlate the differences of gene expression and genetic variations with susceptibility to AS.

DETAILED DESCRIPTION:
This is a matched case-control study to identify genetic susceptibility factors to Ankylosing Spondylitis (AS).

Patients and family controls selected from 154 families have been included in genome-wide linkage screening, comprising 440 patients and 904 individuals genotyped using microarrays Affymetrix® 250,000 single-nucleotide polymorphism (SNPs). For each locus,families with a LOD score of 0;15 in predefined region were retained. In these families will be selected a patient and a healthy control of the same sex, if possible, siblings and of comparable age (<10 years apart).

The patients and controls will be contacted by mail and / or telephone to obtain their participation in this study. An updating Questionnaire of AS events will be sent to them, particularly to check that the family controls did not develop AS since their inclusion in the genetic study.

Patient and family controls recruitment and obtaining their dendritic cells (DC) will be made during the first year.

After signing the informed consent, 60ml of whole blood will be taken from each included subject. The cells obtained from blood samples (leukocytes) will be cultured in the laboratory for seven days and used to extract the RNA that will be used to conduct the research. Some of these cells as well as their RNA will be frozen and can be thawed for later use if required.

Mononuclear cells are isolated from whole blood by gradient centrifugation (Ficoll). CD14 + monocytes will be selected after labeling with an anti-CD14 antibody coupled to ferromagnetic beads (Dynabeads) and the magnet system Dynal, then differentiated in the presence of GM-CSF (Granulocyte Macrophage Colony Stimulating Factor) and IL-4 (Interleukine 4) for 6 days into immature DC (dendritic cells), according to a protocol validated in the laboratory and used in routine. DC maturation is then induced by the addition of lipopolysaccharide E. coli (Sigma) for 18 hours. The pellets of DC will be retained in RNAlater® for extracting RNA.

A transcriptomic study of mature DCs will be carried at the end of the recruitment and will run for two months, including one month of experimentation and 1 month for analysis. This study will be performed using microarrays of genome-wide exon-centric expression. The analyzes will be performed separately for each locus of interest and will bear on the expression of genes localized in each region. The level of transcripts will be normalized for patients and family controls compared to that of a group of 15 controls from the general population already obtained. For each locus, genes having statistically different expression between the group of patients and the family controls and a differential expression ≥ 1 will be identified. The expression level of these genes will then be verified by quantitative real-time PCR (polymerase chain reaction).

The positional and functional candidate genes identified due to a differential expression of their transcripts will be fully re-sequenced to search for polymorphisms that may be responsible for a change in their level of expression.

The investigators expect to study one to three genes per region. The re-sequencing will be performed primarily in patients and family controls with a different level of expression of these genes. Polymorphisms distributed differently between these two populations will be retained for the rest of the study.

The re-sequencing of these candidate genes will be spread over a period of 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient >18 and
* Axial SpA patients fulfilling the ASAS criteria (31) and belonging to families already included in genetic analyses previously made by our Consortium.
* Family controls without AS and matched to AS cases on age, sex and HLA-B27 positivity.
* Non-family independent healthy controls
* Written informed consent

Exclusion Criteria:

* Person specially Protected
* Persons living abroad, in the DOM-TOM

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Ankylosing Spondylitis (AS) and matched family controls from families having a LOD score ≥ 0.15.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2011-08; Primary Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Comparison of the transcriptome of dendritic cells derived from circulating monocytes between cases and controls | 18 months

SECONDARY OUTCOMES:
Assessment of manifestations of Ankylosing Spondylitis (AS) according an Updating Questionnaire. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Maxime BREBAN, MD, PhD, Principal Investigator — Ambroise Paré Hospital, 92100 Boulogne-Billancourt, France
Locations (1):
- Ambroise Paré Hospital, Boulogne-Billancourt, Hauts-De-Seine, France